CLINICAL TRIAL: NCT07285369
Title: Ambroxol in Type III Gaucher Disease (GD3): A Prospective 6-Month Single-Center Open-Label Study With an Optional 12-month Extension Phase
Brief Title: High-Dose Ambroxol in Pediatric Type III Gaucher Disease (GD3)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Agyany Pharma LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGP3
Record Dates: First submitted 2025-11-21; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Gaucher Disease, Type 3
Keywords: Type III Gaucher Disease; Gaucher Disease; GD3; Ambroxol; Pharmacologic chaperone; Ataxia; Myoclonus; Neurological manifestations; Lysosomal storage disorder
MeSH Terms: conditions — Gaucher Disease; Ataxia; Myoclonus; Neurologic Manifestations; Lysosomal Storage Diseases | interventions — Ambroxol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-Dose Ambroxol (Experimental): All participants will receive high-dose Ambroxol orally at a mean dose of 35 mg/kg bodyweight daily for 6 months, with an optional 12-month extension. The drug may be administered with or without enzyme replacement therapy (ERT).
  Interventions: Drug: Ambroxol

INTERVENTIONS:
Drug: Ambroxol — High-dose Ambroxol will be administered orally at a mean dose of 35 mg/kg bodyweight daily. Participants will receive treatment for 6 months, with an optional 12-month extension. The drug may be given with or without concurrent enzyme replacement therapy (ERT).

SUMMARY:
Type: Prospective, open-label, single center study

Duration: 6 months with an optional 12-month extension phase

Participants: 12 pediatric patients diagnosed with type III Gaucher disease (GD3) aged ≥3 to ≤18 years old treatment naïve or on enzyme replacement therapy (ERT). They will be treated with high-dose Ambroxol (mean 35mg/kg bodyweight).

Location: The Children's Hospital, Lahore, Pakistan.

DETAILED DESCRIPTION:
This single-center, prospective, open-label study investigates the safety, tolerability, and efficacy of high-dose Ambroxol in pediatric patients with genetically confirmed Type III Gaucher Disease (GD3). The study will enroll 12 participants aged 3 to 18 years, either treatment naïve or receiving enzyme replacement therapy (ERT). Participants will receive high-dose Ambroxol orally (mean 35 mg/kg bodyweight) over a 6-month period, with an optional 12-month extension.

Primary Objective:

Evaluate the safety and tolerability of high-dose Ambroxol administered with or without ERT.

Secondary Objective:

Assess efficacy based on at least a 20% improvement in at least 50% of participants using the following measures:

* Assessment and Rating of Ataxia (SARA) for patients with ataxia
* Unified Myoclonus Rating Scale (UMRS) for patients with myoclonic epilepsy
* Lyso-Gb1 levels in peripheral blood after at least 6 months of treatment

Intervention:

High-dose Ambroxol administered orally (mean 35 mg/kg bodyweight)

Study Location:

The Children's Hospital, Lahore, Pakistan

This study aims to provide preliminary safety and efficacy data on Ambroxol as a therapeutic option for pediatric patients with GD3, potentially informing future larger-scale clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 3 to 18 years
* Genetically confirmed Type III Gaucher Disease (GD3)
* Treatment naïve or receiving enzyme replacement therapy (ERT)
* SARA score ≥ 8
* Sexually active females must agree to use contraception
* All participants must not be pregnant or breastfeeding

Exclusion Criteria:

* Life-threatening visceral disease (related or unrelated to Gaucher Disease)
* Blood transfusion dependency
* Clinically significant cardiovascular, gastrointestinal, pulmonary, neurologic, endocrine, or psychiatric conditions
* Serious swallowing difficulties
* Renal insufficiency (eGFR < 30 mL/min/1.73 m²)
* Recent chaperone therapy or investigational treatment within the last 6 months
* Pregnancy or lactation
* History of cancer, drug or alcohol abuse, major organ transplant, or inability to adhere to study requirements

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of High-Dose Ambroxol | 6 months (with optional assessment at 12-month extension)
  Incidence and Severity of Treatment-Emergent Adverse Events

SECONDARY OUTCOMES:
Assess the efficacy of high-dose (mean 35mg/kg bodyweight) Ambroxol by at least 20% improvement in at least 50% of the patients measured with: assessment and Rating of Ataxia (SARA) scale for patients with ataxia. | 6 months (with optional assessment at 12-month extension)
  50% of Participants Achieving ≥20% Improvement in SARA Score

CONTACTS AND LOCATIONS:
Overall Officials: Huma Arshad Cheema, Prof., Principal Investigator — The Children's Hospital, Lahore, Pakistan
Locations (1):
- The Children's Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided